CLINICAL TRIAL: NCT05331755
Title: Real Life Experience Survey of Dupilumab in the Netherlands
Acronym: RELYonDupi
Status: Completed | Type: Observational
Sponsor: Gert-Jan Braunstahl (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor-Investigator, Gert-Jan Braunstahl, Principal Investigator, Franciscus Gasthuis
Organization: Franciscus Gasthuis (Other)
Other Study IDs: SGZ-2021-13401
Record Dates: First submitted 2022-04-02; First posted 2022-04-18 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Severe Asthma
MeSH Terms: conditions — Asthma | interventions — dupilumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Severe T2 high asthma: Included patients will have severe type 2 high asthma, are eligible for dupilumab conform EU label, minimally treated with high dose ICS and LABA and have:
  * blood eosinophils 150 - 1500/mm2 OR
  * FeNO >20 ppb OR
  * clinical significant inhalation allergy (+ sIgE positive) OR
  * OCS dependency
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab — start medication in cohort
  Other Names: Dupixent

SUMMARY:
Rationale: Dupilumab has proven to be effective and safe in several large randomized controlled trials. However, study populations in RCT's represent only a small proportion of severe asthma patients treated in real life circumstances. Therefore, real-life studies provide data complementary to RCT's derived from a more diverse and heterogeneous group of patients. This study is unique in that it represents a large population of European patients that are not represented in the Global Registry.

Objective: To collect and analyse efficacy and safety data in severe asthma patients treated with dupilumab in a real-life setting.

Study design: Single center, retrospective cohort analysis of severe asthma patients treated with dupilumab, as decided by the treating physician.

Setting: Severe Asthma Expert Center Franciscus Gasthuis & Vlietland, Rotterdam Study population: All patients that started with dupilumab from jan 2019 (early access program) until June 2020 are eligible for the study. They should be 18 years or older, with severe T2 high asthma and treated with at least one dose of dupilumab.

Main study parameters/endpoints:

* Primary endpoint: To assess changes in annual exacerbation rate between baseline and after 12 months treatment in severe asthma patients treated with dupilumab.
* Secondary endpoints: To collect data on ACQ, OCS use, FEV1, treatment response rate, influence of co-morbidities and safety.

Methods:

Exacerbation history and patient characterization will be done at baseline. We aim to include patients in the analysis that had at least one administration of dupilumab (intention-to-treat). Treatment response evaluation is done at 12 months. Final evaluation of efficacy and safety is done at 12 months of treatment. We aim to enroll at least 120 patients in the study. Data collection will be done in Castor Electronic Data Capture. Of the 120 patients scheduled for inclusion, all have already started treatment and data will be collected retrospectively at the predefined time points. Patient data will be handled confidentially.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Since this is a retrospective cohort analysis there are no extra visits, interventions or procedures needed. Therefore, there is no increased burden or risk for the patients involved.

DETAILED DESCRIPTION:
1. INTRODUCTION AND RATIONALE

   Background:

   Severe asthma is a rare condition affecting approximately 5% of all asthma patients. Patients experience daily symptoms and often have frequent exacerbations despite the use of high dose ICS and LABA. Influencing factors such as co-morbidity and non-adherence to therapy are optimized. Nevertheless, they continue having uncontrolled asthma or can only be controlled with systemic corticosteroids.

   Dupilumab is a monoclonal anti-IL-4Rα antibody developed for the treatment of severe asthma. It effectively targets both the IL-4 and IL-13 pathway, resulting in reduction of asthma exacerbations and improvement of asthma control in patients with T2-high asthma. T2-inflammation is defined by the presence of eosinophils in sputum or blood, clinically relevant allergic sensitization and/or increased fraction of exhaled nitric oxide (FeNO). This type of inflammation is present in 60-70% of severe asthma patients. Severe asthma is a heterogeneous group of asthma phenotypes which are not all represented well in previously performed clinical trials. Therefore, it is of importance to conduct real-life studies which include all kind of patients regardless of co-morbidity, environmental exposures, previous treatment with biologicals or ethnical background. These studies provide the necessary data that complement to those obtained by RCT's.

   To date, little is known about the response rate, efficacy, and safety of dupilumab in daily practice. To our knowledge, this study will be the largest study to date to assess response rate, efficacy as well as safety in patients with severe T2-high asthma who are treated with at least one dose of dupilumab. The investigators expect 80% of the patients to respond to dupilumab. This is in line with the French cohort of dupilumab in real life published bij Dupin et al. Furthermore, half of the patients will be on chronic OCS treatment, these patients are expected to respond well, even so patients with nasal polyposis and atopic eczema. The investigators expect a reduction in mean ACQ of 0.8 point (MCID = -0,5) and in asthma-exacerbations of at least 70% compared to baseline (MCID = -30%). This would be in line with previous real life biological studies that the investigators performed in and the French cohort. As for post-FEV1 the investigators expect an increase of 10% predicted during the study period. The investigators expect 40% to be super-responders.

   Study rationale:

   Dupilumab has proven to be effective and safe in several large randomized controlled trials. However, study populations in RCT's represent only a small proportion of severe asthma patients treated in real life circumstances. Therefore, real-life studies provide data complementary to RCT's derived from a more diverse and heterogeneous group of patients.
2. OBJECTIVES

   Primary objectives:

   To assess changes in annual exacerbation rate prior to and after 12 months treatment in severe asthma patients treated with dupilumab.

   Secondary objectives:
   * Patient characterization, including severity and inflammatory profile,
   * Diagnosis and referral history,
   * Responder rate and average treatment time with dupilumab,
   * Efficacy in patients previously treated with biologicals (anti-IgE, anti-IL5),
   * Change in lung function,
   * Change in asthma control,
   * Reduction of comedication,
   * Reduction in hospital admissions
   * Effect on comorbidities,
   * Safety issues.
3. STUDY DESIGN Single center, retrospective cohort analysis of severe asthma patients treated with dupilumab, as decided by the treating physician. The follow-up period is one-year after start of therapy. Patients that stopped treatment with dupilumab during the follow-up year are also included in the data analysis.
4. STUDY POPULATION 4.1 Population (base)

   Included patients will have severe type 2 high asthma, are eligible for dupilumab conform EU label, minimally treated with high dose ICS and LABA and have:
   * blood eosinophils 150 - 1500/mm2 OR
   * FeNO >20 ppb OR
   * clinical significant inhalation allergy (+ sIgE positive) OR
   * OCS dependency

   The investigators have access to dupilumab since January 2019 (early access program); from June 2019 on dupilumab was registered in the Netherlands. To date, the investigators have 143 patients on dupilumab treatment. There is no extra burden for the patient because there is no intervention and because the visits and outcome parameters described in this proposal are already part of standard care in the Institution, a tertiary referral centre. Therefore, the investigators expect to include at least 85% of the patients. Our back-up plan is to extend the study to our regional severe asthma network South-West Netherlands, which comprises 11 general hospitals and 1 academic centre.

   4.2 Inclusion criteria All patients that started with dupilumab from Jan 2019 (early access program) until June 2020 are eligible for the study. They should be 18 years or older, with severe T2 high asthma and treated with at least one dose of dupilumab. All included patients should provide written informed consent.

   4.3 Exclusion criteria Patients with COPD (Chronic Obstructive Pulmonary Disease) or EGPA (Eosinophilic Granulomatosis with PolyAngiitis) will be excluded.

   Also, patients that had dupilumab prescribed for other reasons (nasal polyposis or atopic dermatitis) will be excluded as well.

   4.4 Sample size calculation Since the study is retrospective and observational in nature, no sample size calculation needs to be done.
5. TREATMENT OF SUBJECTS Patients will be uploaded with 600 mg when having atopic eczema or nasal polyposis as a co-morbid condition next to their severe asthma or when on maintenance treatment with OCS. In all other cases 400 mg dupilumab was considered sufficient. After the first dose treatment was continued with resp. 300 mg or 200 mg according to the local protocol. The first three injections were given in the hospital. After the third injection patients were allowed to proceed with self-injection at home. During the first year of treatment patients were followed-up at regular intervals either by outpatient visit or telephone call.

   5.1 Summary of findings from non-clinical studies Dupilumab is a monoclonal anti-IL-4Rα antibody developed for the treatment of severe asthma. It effectively targets both the IL-4 and IL-13 pathway.

   5.2 Summary of findings from clinical studies Treatment with dupilumab results in reduction of asthma exacerbations and improvement of asthma control in patients with T2-high asthma.

   5.3 Summary of known and potential risks and benefits Dupilumab is already registered for the treatment of severe T2-high asthma. It has proven to be effective and safe in RCT's. However, it is of importance to conduct real-life studies which include all kind of patients regardless of co-morbidity, environmental exposures, previous treatment with biologicals or ethnical background. These studies provide the necessary data that complement to those obtained by RCT's.
6. METHODS 6.1 Study parameters/endpoints 6.1.1 Main study parameter/endpoint To assess asthma exacerbation* rate annually at both baseline (up to 12 months prior to the start of dupilumab therapy) and after 12 months of dupilumab therapy.

   6.1.2 Secondary study parameters/endpoints (if applicable)
   * Patient characterization, including severity (GINA score), Medical Research Council- dyspnea scale (MRC), FeNO (ppb) and blood eosinophils (abs nr).
   * Diagnosis and referral history, including time between diagnosis, referral and treatment initiation.
   * Responder rate, according to predefined criteria** (super response, partial response and no response).
   * Average treatment time with dupilumab after 12 months follow-up (total group).
   * Exacerbation rate at 6 months.
   * Change in asthma control*** (ACQ-5)
   * Efficacy in patients previously treated with biologicals (anti-IgE, anti-IL5).
   * Change in lung function (FEV1) in mL and %pred; change in FeNO (ppb).
   * Reduction of comedication, including dose of oral corticosteroids (OCS).
   * Hospital admission; historical data 1 year before start until 1 year after start of dupi-lumab.
   * Effect on comorbidities, including atopic dermatitis, sinusitis and nasal polyps.
   * Safety, adverse events and serious adverse events (aligning with Sanofi require-ments).

     * Asthma exacerbation: increase of asthma symptoms above daily variation requiring treatment with oral corticosteroids for at least 3 days.

       * Super responders were defined as follows: meeting at least 3 or more criteria (2 of which should be major) and should be assessed over 12 months.

   Major criteria:
   * No exacerbations
   * Major improvement in asthma control (2x MCID)
   * No maintenance OCS (or weaning to adrenal insufficiency)

   Minor Criteria:
   * 75% exacerbation reduction
   * Well-controlled asthma (ACQ < 1.0)
   * More than 500 mL improvement in FEV1

   Patients were considered partial responders after 12 months when they met at least 1 (but < 3) of the above-mentioned criteria after 12 months of dupilumab therapy.

   Non-responders were characterized by meeting none of the above criteria and/or quitting dupilumab before 12 months due to insufficient efficacy according to the treating physician or patient.

   *** Asthma control, using Asthma Control Questionnaire (ACQ, Juniper 1999): the investigators use the ACQ-5 comprising 5 questions about symptoms. An improvement of 0,5 is considered to be clinically significant.

   6.2 Randomisation, blinding and treatment allocation NA

   6.3 Study procedures Data were collected from the digital patient file system of the Sint Franciscus Hospital Rotterdam (HiX: Healthcare Information eXchange, Chipsoft BV, Amsterdam, The Netherlands) and stored in Castor EDC (Castor Electronic Data Capture, Ciwit BV, Amsterdam, The Netherlands).

   Of the 120 patients scheduled for inclusion, all have already started treatment and data will be collected retrospectively at the predefined time points: At start of dupilumab therapy (baseline), at 6 months- and at 12 months after initiation of dupilumab therapy. Patient data will be handled confidentially. For each subject a unique identification code will be used to link the data to the subject. The personal data will be handled according to the General Data Protection Regulation (GDPR). Patients will be asked for written informed consent to share their clinical information anonymously.

   6.4 Withdrawal of individual subjects All patients will be asked for their consent prior to data collection. Subjects can withdraw their consent at any time for any reason if they wish to do so without any consequences.

   6.5 Replacement of individual subjects after withdrawal NA

   6.6 Follow-up of subjects withdrawn from treatment Patients that stopped with dupilumab within one year after start of the treatment will be included in the data analysis following the intention-to-treat principle.

   6.7 Premature termination of the study NA
7. SAFETY REPORTING 7.1 Temporary halt for reasons of subject safety NA

   7.2 AEs, SAEs and SUSARs 7.2.1 Adverse events (AEs) Adverse events are defined as any undesirable experience occurring to a subject during the study, whether or not considered related to [the investigational product / trial procedure/ the experimental intervention]. All adverse events reported spontaneously by the subject or observed by the investiga¬tor or his staff will be recorded.

   7.2.2 Serious adverse events (SAEs) A serious adverse event is any untoward medical occurrence or effect that
   * results in death;
   * is life threatening (at the time of the event);
   * requires hospitalisation or prolongation of existing inpatients' hospitalisation;
   * results in persistent or significant disability or incapacity;
   * is a congenital anomaly or birth defect; or
   * any other important medical event that did not result in any of the outcomes listed above due to medical or surgical intervention but could have been based upon appropriate judgement by the investigator.

   An elective hospital admission will not be considered as a serious adverse event.

   7.2.3 Suspected unexpected serious adverse reactions (SUSARs) NA

   7.3 Annual safety report NA
8. STATISTICAL ANALYSIS 8.1 Primary study parameter(s) The primary effectiveness analysis will be performed on the intent-to-treat (ITT) population comparing exacerbation rate at 12 months after first dose of dupilumab with exacerbation rate in the year prior to initiation. The ITT population comprises all enrolled patients who received at least one dose of dupilumab and had at least one post-baseline effectiveness assessment.

   8.2 Secondary study parameter(s) Demographic and other baseline characteristics will be summarized using descriptive statistics. All results are expressed as median for continuous variables, and number (%) for categorical variables. Efficacy tables will also be created for the per protocol (PP) population to measure the impact on the results of patients with at least one major protocol deviation. The safety population comprises all patients who were enrolled in the database, who received at least one dose of dupilumab and had at least one post-baseline safety assessment. Descriptive summaries are presented for treatment effect, asthma exacerbations, FEV1, ACQ-5, eosinophils, FeNO, hospitalizations and OCS use.

   Subgroup analysis will be done with the binomial regression model. Subgroup analyses will be conducted on 3 predefined endpoints: previous biological use, atopy and nasal polyps. Each subgroup will be evaluated for treatment response, ACQ, FEV1 (mL), FEV1 (%) predicted, use of OCS and OCS dose at 12 months. The investigators will compare the outcomes with historical data in the literature for magnitude of clinical effect. No direct comparisons will be made. Data analysis will be performed with SPSS statistics version 27 (IBM SPSS).

   8.3 Interim analysis (if applicable) NA
9. ETHICAL CONSIDERATIONS 9.1 Regulation statement The personal data will be handled according to the General Data Protection Regulation (GDPR).

   9.2 Recruitment and consent Patient data will be handled confidentially. For each subject a unique identification code will be used to link the data to the subject. Patients will be asked for written informed consent to share their clinical information anonymously.

   9.3 Objection by minors or incapacitated subjects (if applicable) NA

   9.4 Benefits and risks assessment, group relatedness Dupilumab is already registered for the treatment of severe T2-high asthma. It has proven to be effective and safe in RCT's. However, it is of importance to conduct real-life studies which include all kind of patients regardless of co-morbidity, environmental exposures, previous treatment with biologicals or ethnical background. These studies provide the necessary data that complement to those obtained by RCT's.

   9.5 Compensation for injury NA

   9.6 Incentives (if applicable) NA
10. ADMINISTRATIVE ASPECTS, MONITORING AND PUBLICATION 10.1 Handling and storage of data and documents Data collection will be done in Castor Electronic Data Capture. Of the 120 patients scheduled for inclusion, all have already started treatment and data will be collected retrospectively at the predefined time points. Patient data will be handled confidentially. For each subject a unique identification code will be used to link the data to the subject. The personal data will be handled according to the General Data Protection Regulation (GDPR). Patients will be asked for written informed consent to share their clinical information anonymously.

10.2 Monitoring and Quality Assurance An independent monitor (quality officer), appointed by the sponsor, will monitor the study data according to Good Clinical Practice (GCP). The frequency of the monitoring is related to the risk of the investigation. For at least a selection of the subjects, Informed Consents will be checked. Source Data Verification will not or minimally be performed (checking if data from the Case Report Forms (research forms / questionnaires) matches with the source data (patient status, results, etc.)). The quality of data will be guaranteed by using the data management software Castor EDC. The monitor will check whether all (S)AEs and SUSARs are adequately reported within the timelines as required by law, the presence and correctness of the Informed consent forms, the delegation log and the data storage

10.3 Amendments All substantial amendments will be notified to the METC and to the competent authority.

Non-substantial amendments will not be notified to the accredited METC and the competent authority but will be recorded and filed by the sponsor.

10.4 Annual progress report The sponsor/investigator will submit a summary of the progress of the trial to the accredited METC once a year. Information will be provided on the date of inclusion of the first subject, numbers of subjects included and numbers of subjects that have completed the trial, serious adverse events/ serious adverse reactions, other problems, and amendments.

10.5 Temporary halt and (prematurely) end of study report The investigator/sponsor will notify the accredited METC of the end of the study within a period of 8 weeks. The end of the study is defined as the last patient's included in the data file.

The sponsor will notify the METC immediately of a temporary halt of the study, including the reason of such an action.

In case the study is ended prematurely, the sponsor will notify the accredited METC within 15 days, including the reasons for the premature termination.

Within one year after the end of the study, the investigator/sponsor will submit a final study report with the results of the study, including any publications/abstracts of the study, to the accredited METC.

10.6 Public disclosure and publication policy Data will be disclosed after review by sponsor/PI and published on conferences and medical journals.

ELIGIBILITY:
Inclusion Criteria:

* All patients that started with dupilumab from Jan 2019 (early access program) until June 2020 are eligible for the study. They should be 18 years or older, with severe T2 high asthma and treated with at least one dose of dupilumab. All included patients should provide written informed consent.

Exclusion Criteria:

* Patients with COPD (Chronic Obstructive Pulmonary Disease) or EGPA (Eosinophilic Granulomatosis with PolyAngiitis) will be excluded.

Also, patients that had dupilumab prescribed for other reasons (nasal polyposis or atopic dermatitis) will be excluded as well.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Included patients will have severe type 2 high asthma, are eligible for dupilumab conform EU label, minimally treated with high dose ICS and LABA and have:
  * blood eosinophils 150 - 1500/mm2 OR
  * FeNO >20 ppb OR
  * clinical significant inhalation allergy (+ sIgE positive) OR
  * OCS dependency
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Annual exacerbation rate | 12 months before and after start medication
  To assess changes in annual exacerbation rate prior to and after 12 months treatment in severe asthma patients treated with dupilumab.

SECONDARY OUTCOMES:
Change in lung function | 12 months before and after start medication
  FEV1
Change in asthma control | 12 months before and after start medication
  ACQ

OTHER OUTCOMES:
% of patients with atopy | 12 months before and after start medication
  positive inhalation screen (Phadiatop)
% patients referred from other hospitals | 12 months before and after start medication
  percentage
Responder rate and average treatment time with dupilumab | 12 months before and after start medication
  percentage responders and months treated with dupilumab
Efficacy in patients previously treated with biologicals (anti-IgE, anti-IL5) | 12 months before and after start medication
  change in biological switchers
Change in co-medication | 12 months before and after start medication
  change in dose of LABA, LAMA, ICS, OCS
Reduction in hospital admissions | 12 months before and after start medication
  number of hospital admissions
Percentage of patients with relevant co-morbidities | 12 months before and after start medication
  Percentage of patients with nasal polyps, atopic dermatitis
Percentage of patients with safety issues | 12 months before and after start medication
  percentage and classification of AE, SAE

CONTACTS AND LOCATIONS:
Overall Officials: Jursica Mills, MSc, Study Director — Wetenschapsbureau FGV
Locations (1):
- Franciscus Gasthuis & Vlietland, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Our data will be available to anyone upon request

REFERENCES:
- [Background] 4. Update asthma guidelines 2020 (Global Initiative for Asthma): www.ginasthma.org.
- [Background] Dupin C, Belhadi D, Guilleminault L, Gamez AS, Berger P, De Blay F, Bonniaud P, Leroyer C, Mahay G, Girodet PO, Raherison C, Fry S, Le Bourdelles G, Proust A, Rosencher L, Garcia G, Bourdin A, Chenivesse C, Didier A, Couffignal C, Taille C. Effectiveness and safety of dupilumab for the treatment of severe asthma in a real-life French multi-centre adult cohort. Clin Exp Allergy. 2020 Jul;50(7):789-798. doi: 10.1111/cea.13614. Epub 2020 May 29. PMID 32469092
- [Result] Hekking PW, Wener RR, Amelink M, Zwinderman AH, Bouvy ML, Bel EH. The prevalence of severe refractory asthma. J Allergy Clin Immunol. 2015 Apr;135(4):896-902. doi: 10.1016/j.jaci.2014.08.042. Epub 2014 Oct 16. PMID 25441637
- [Result] Rabe KF, Nair P, Brusselle G, Maspero JF, Castro M, Sher L, Zhu H, Hamilton JD, Swanson BN, Khan A, Chao J, Staudinger H, Pirozzi G, Antoni C, Amin N, Ruddy M, Akinlade B, Graham NMH, Stahl N, Yancopoulos GD, Teper A. Efficacy and Safety of Dupilumab in Glucocorticoid-Dependent Severe Asthma. N Engl J Med. 2018 Jun 28;378(26):2475-2485. doi: 10.1056/NEJMoa1804093. Epub 2018 May 21. PMID 29782224
- [Result] Castro M, Corren J, Pavord ID, Maspero J, Wenzel S, Rabe KF, Busse WW, Ford L, Sher L, FitzGerald JM, Katelaris C, Tohda Y, Zhang B, Staudinger H, Pirozzi G, Amin N, Ruddy M, Akinlade B, Khan A, Chao J, Martincova R, Graham NMH, Hamilton JD, Swanson BN, Stahl N, Yancopoulos GD, Teper A. Dupilumab Efficacy and Safety in Moderate-to-Severe Uncontrolled Asthma. N Engl J Med. 2018 Jun 28;378(26):2486-2496. doi: 10.1056/NEJMoa1804092. Epub 2018 May 21. PMID 29782217
- [Result] Snelder SM, Weersink EJM, Braunstahl GJ. 4-month omalizumab efficacy outcomes for severe allergic asthma: the Dutch National Omalizumab in Asthma Registry. Allergy Asthma Clin Immunol. 2017 Jul 26;13:34. doi: 10.1186/s13223-017-0206-9. eCollection 2017. PMID 28769983
- [Result] van Toor JJ, van der Mark SC, Kappen JH, In 't Veen JCCM, Braunstahl GJ. Mepolizumab add-on therapy in a real world cohort of patients with severe eosinophilic asthma: response rate, effectiveness, and safety. J Asthma. 2021 May;58(5):651-658. doi: 10.1080/02770903.2020.1723623. Epub 2020 Feb 12. PMID 31999203
- [Result] Upham JW, Le Lievre C, Jackson DJ, Masoli M, Wechsler ME, Price DB; Delphi Panel. Defining a Severe Asthma Super-Responder: Findings from a Delphi Process. J Allergy Clin Immunol Pract. 2021 Nov;9(11):3997-4004. doi: 10.1016/j.jaip.2021.06.041. Epub 2021 Jul 13. PMID 34271216